CLINICAL TRIAL: NCT06697249
Title: Feasibility of Valve-in-Root Transcatheter Aortic Valve Implantation in 363 Patients After Aortic Root Replacement and Repair: a Retrospective Computed-tomography Analysis
Brief Title: Feasibility of Valve-in-Root Transcatheter Aortic Valve Implantation in 363 Patients After Aortic Root Replacement and Repair
Acronym: Valve in Root
Status: Completed | Type: Observational
Sponsor: Alicja Zientara (Other)
Responsible Party: Sponsor-Investigator, Alicja Zientara, Principal investigator, University Hospital Freiburg
Organization: University Hospital Freiburg (Other)
Other Study IDs: ViR 2024
Record Dates: First submitted 2024-10-02; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Aortic Valve Disease Mixed; Transcatheter Aortic Valve Replacement
Keywords: Valve-in-root aortic valve replacement; transcatheter aortic valve replacement; root replacement; valve-sparing aortic root replacement

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- RR patients: Patients after biological aortic root replacement
  Interventions: Other: Analysis of postoperative CT scans checking for the feasibility of transcatheter valve-in-root implantation
- VSRR patients: Patients after valve-sparing aortic root replacement
  Interventions: Other: Analysis of postoperative CT scans checking for the feasibility of transcatheter valve-in-root implantation

INTERVENTIONS:
Other: Analysis of postoperative CT scans checking for the feasibility of transcatheter valve-in-root implantation — CT scans of patients after biological root replacement and root repair were assessed with the 3mensio Software (Aortic valve package, 3mensio 10.1, Pie Medical Imaging. Before carrying out the measurements, markers for alignment of the aortic root and ascending aorta were placed manually. The annular area was measured for both groups. In patients after biological root replacement the area of the annulus was defined as the ring of the initial aortic valve prosthesis. Coronary buttons were measured at their lowest and highest point to define partial or full position below the valve level and the general button size. For assessment of the annular-to-coronary distance, the lower edge of the coronary button was chosen. VTC was assessed after root replacement in patients who had at least one coronary partially under the level of the valve. For this measurement a virtually inserted valve was placed in the bioprosthetic frame.

SUMMARY:
Biological replacement of the aortic valve in the sense of a complete root replacement is the therapy for a dilatation or aneurysm of the ascending aorta, which also involves the aortic valve. In some patients, the aortic valve can be preserved, which means that only reconstruction is necessary instead of a complete replacement of the root. For a root replacement or root reconstruction, both coronary arteries must be prepared at their origin from the aorta and reimplanted into a tubular prosthesis. It is known that biological aortic valve prostheses have a lifespan of between 10-20 years depending on the type and design of the valve and that the first degenerative symptoms become visible after 10-12 years. This is particularly relevant for patients who have their initial operation at a younger age and require a follow-up procedure if the valve degenerates at an older age.

The minimally invasive implantation of transcatheter valves has proven to be a successful method, avoiding a second operation with an increased risk of mortality. The so-called valve-in-valve procedures are carried out particularly in older patients and are now standard in modern valve treatment. The feasibility of a valve-in-valve in the aortic position requires certain anatomical conditions, which can be influenced by the surgeon's implantation technique in the case of additional root replacement. In particular, there is a risk of coronary artery occlusion when implanting the transcatheter valve, which is increased if the coronary artery branches are located below the valve level. In addition, the selection of the prosthesis size is an important parameter for subsequently implanting a suitably large transcatheter valve.

The aim of this study is to use postoperative computer tomography of patients after root replacement/reconstruction to measure the anatomical parameters that describe a possible implantation of a transcatheter valve in the event of degeneration of the initial valve. This simultaneously shows the quality of the root replacement/reconstruction with regard to a plannable follow-up procedure and can also show for the future how the surgical technique could be modified to make a minimally invasive follow-up intervention available to more patients.

This study aims to answer the question of whether the patients who were treated with biological root replacement or reconstruction in the years 2012-2022 for aortic valve failure are anatomically suitable for valve-in-valve therapy based on the postoperative computed tomography measurements of the aortic root. In addition, the measurements provide a surgical answer to the question of whether relevant parameters such as the distance between the coronary arteries were sufficiently taken into account during the initial operation or whether an improvement should be made in the future while adhering to the anatomically important parameters during the initial procedure.

ELIGIBILITY:
Inclusion Criteria:

* all patients over 18 years after biological aortic root replacement or repair
* postoperative ECG-gated CT-angiography scan

Exclusion Criteria:

* mechanical aortic root replacements (not suitable for Valve-in-Root treatment)
* missing postoperative ECG-gated CT-angiography scan

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From January 2012 till December 2022, 760 patients underwent either an aortic root replacement or valve-sparing root replacement using the David technique. All patients over the age of 18 were included. The exclusion criteria were mechanical aortic root replacements and a missing postoperative ECG-gated CT-angiography scan of the thoracic aorta resulting in cumulatively 363 patients after either biological root replacement or root repair. The CT scans were obtained before discharge or during the first two years after the operation in the context of the routine postoperative follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 760 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
CT-measurement: Aortic annulus area | January 2024-June 2024
CT-measurement: Valve-to-coronary distance | January 2024-June 2024
CT measurement: Annulus-to-coronary distance | January 2024-June 2024
CT-measurement: Size of coronary buttons | January 2024-June 2024

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital Freiburg, Department of Cardiovascular Surgery, Freiburg im Breisgau, Germany

IPD SHARING:
Plan to Share IPD: No